CLINICAL TRIAL: NCT01203761
Title: The Experience of Loneliness Among Ear, Nose and Throat (ENT) Surgical Patients During the Perioperative Period
Brief Title: The Experience of Loneliness Among Patients During the Perioperative Period
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Professor Idit Matot. Chair, Department of Anesthsiology & Intensive Care, Tel-Aviv Sourasky Medical Center
Other Study IDs: TASMC-10-IM-0301-CTIL
Record Dates: First submitted 2010-09-01; First posted 2010-09-16 (Estimated); Last update posted 2010-09-16 (Estimated); Status verified 2010-09

CONDITIONS: Anxiety; Depression
Keywords: loneliness
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Preoperative patients: ENT surgical patients, approximately 1 day before their procedure undertaken
- Postoperative patients: ENT surgical patients during their postoperative hospitalization
- Family members: Family members of ENT surgical patients, during the perioperative period

SUMMARY:
The experience of illness and hospitalization exerts a great deal of psychological distress, one of the most distressful events people might experience throughout their life times. Surgery and anesthesia with their accompanying loss of control, fear of being unconscious and invaded, and expectation of postoperative pain adds appreciably to that stress and anxiety.

Current psycho-physiological research has provided evidence on the alarming possibility of the aversive affects of hospitalization stress on the patients' already deteriorated physical health and marked interference with their recovery.

As an additional stressor, which may partly be related to the hospital staff, and partly to the person's illness and expected surgery is loneliness.

Loneliness is a painful experience that is, commonly, not embraced and which has consequences that are detrimental to one's emotional, physical and spiritual well being.

The present study explores the qualitative aspects of loneliness (via questionnaires) in two patient populations: (1) patients facing surgery, and (2) patients who have already undergone surgery. In addition, family members [i.e. those waiting outside of the operating room] will be given a questionnaire, and these three groups will be compared to the general population.

DETAILED DESCRIPTION:
The modern hospital environment is generally perceived to provide a safe and healing environment for people inflicted with a variety of illnesses, be it for short term visits and minor health problems or more serious conditions requiring long term treatment and care. However, the experience of illness and hospitalization nonetheless exerts a great deal of psychological distress, one of the most distressful events people might actually experience in their life time [1].

From the outset, illness itself is a major stressor on one's life. However, surgery, with its accompanying loss of control, fear of being invaded, and expectation of post operative pain adds appreciably to that stress and anxiety. Current psycho-physiological research has provided evidence on the alarming possibility of the aversive affects of hospitalization stress on the patients' already deteriorated physical health and marked interference with their recovery [1].

Despite the best intentions of most hospital staffs, emotional distance and depersonalization of the patients might be their natural reaction in dealing with the harsh reality of the patients' ill fate and enormous demands of their responsibilities without being burned out or losing their focus of attention on treatment tasks. As an additional stressor, which may partly be related to the hospital staff, and partly to the person's illness and expected surgery is Loneliness.

Loneliness is a painful experience that is, commonly, not embraced and which has consequences that are detrimental to one's emotional, physical and spiritual well being [2,3]. Lonely individuals tend to exhibit negative intrapersonal traits like pessimism [2,4]. Loneliness was found to be negatively correlated with happiness [5] and life satisfaction [6]. It has been linked to such maladies as depression, hostility, alcoholism, poor self-concept, and psychosomatic illnesses [3].

Study design The present study will explore the qualitative aspects of loneliness [not its intensity] in two patient populations: (1) patients facing surgery, and (2) patients who have already undergone surgery. In addition, family members [i.e. those waiting outside of the operating room] will be given a questionnaire, and these three groups will be compared to the general population.

The loneliness questionnaire is a 60 item yes/no questionnaire that will examine the quality of the loneliness that the participant may experience (enclosed with the proposal). Additionally, there will be demographic questions, and information will be sought about the illness of the patient, the number of hospitalization days, and previous hospitalizations or surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Adult (>18 y/o) inpatients of American Society of Anesthesiologists (ASA) I-IV physical statuses, undergoing an elective surgery at the Ear, Nose and Throat (ENT) department of Tel Aviv Sourasky medical center.

Exclusion Criteria:

* Emergency procedures.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population includes 3 groups:
  1. ENT surgical patients in the preoperative period
  2. ENT surgical patients in the postoperative period
  3. Family members of ENT patients, perioperatively
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2010-09; Primary Completion 2011-09 (Estimated); Study Completion 2011-11 (Estimated)

PRIMARY OUTCOMES:
Loneliness | One day before surgery until POD3
  Qualitative evaluation of the loneliness experience

CONTACTS AND LOCATIONS:
Overall Officials: Idit Matot, MD, Study Chair — Tel-Aviv Sourasky Medical Center
Locations (1):
- Tel Aviv Sourasky medical center, Tel Aviv, Israel

REFERENCES:
- [Background] (1) Hughes B. Psychology, hospitalization and some thoughts on medical training. European Journal of Psychotherapy and Counselling 2001;4: 7-26. (2) Ernst JM CJ. Lonely Hearts: Psychological perspectives on loneliness. Applied and Preventative Psychology 1999;8: 1-22. (3) McWhirter B. Loneliness: A review of current literature with implications for counselling and research. Journal of Counselling and Development 1990;68: 417-423. (4) Davis HH, R Edson, C Ziegler. The relationship between optimism-pessimism, loneliness, and levels of self-esteem in college students. College Student Journal 1992;26: 244-247. (5) Booth R BD, Bohnsock J An examination of the relationship between happiness, loneliness, and shy men in college students. Journal of College Student Development 1992;33: 157-162. (6) Riggio RE WK, Throckmorton B. Social skills, social support, and psychosocial adjustment. Personality and Individual Differences 1993;15: 275-308.